CLINICAL TRIAL: NCT05969717
Title: Exploratory Clinical Study on Induced Pluripotent Stem Cell Derived Exosomes (GD-iExo-001) for the Treatment of Atopic Dermatitis
Brief Title: Induced Pluripotent Stem Cell Derived Exosomes for the Treatment of Atopic Dermatitis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Guidon Pharmaceutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K3016
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GD-iExo-001 treatment (Experimental): Group1 (low-dose group), 8 papatients are treated with 10 μg/mL GD-iExo-001. Group2 (high-dose group), 8 papatients are treated with 50 μg/mL GD-iExo-001. One drop (about 50 μL) of GD-iExo-001 was given to the affected skin area of 2-4 cm2 for 14 consecutive days, twice per day.
  Interventions: Drug: GD-iExo-001
- Normal saline control (Placebo Comparator): Group1 (low-dose group), 2 papatients are treated with normal saline. Group2 (high-dose group), 2 papatients are treated with normal saline. One drop (about 50 μL) of normal saline was given to the affected skin area of 2-4 cm2 for 14 consecutive days, twice per day.
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: GD-iExo-001 — One drop (about 50 μL) of GD-iExo-001 was given to the affected skin area of 2-4 cm2 for 14 consecutive days, twice per day.
  Arms: GD-iExo-001 treatment
Other: normal saline — One drop (about 50 μL) of normal saline was given to the affected skin area of 2-4 cm2 for 14 consecutive days, twice per day.
  Arms: Normal saline control

SUMMARY:
Evaluate the safety, tolerability, and preliminary efficacy of GD-iExo-001 in the treatment of atopic dermatitis

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic inflammatory skin disease that is characterised by intense itching and recurrent eczematous lesions. Although it most often starts in infancy and affects two of ten children, it is also highly prevalent in adults. It is the leading non-fatal health burden attributable to skin diseases, inflicts a substantial psychosocial burden on patients and their relatives, and increases the risk of food allergy, asthma, allergic rhinitis, other immune-mediated inflammatory diseases, and mental health disorders. Originally regarded as a childhood disorder mediated by an imbalance towards a T-helper-2 response and exaggerated IgE responses to allergens, it is now recognised as a lifelong disposition with variable clinical manifestations and expressivity, in which defects of the epidermal barrier are central. Present prevention and treatment focus on restoration of epidermal barrier function, which is best achieved through the use of emollients. Topical corticosteroids are still the first-line therapy for acute flares, but they are also used proactively along with topical calcineurin inhibitors to maintain remission.

Exosomes are nano-sized biovesicles released into surrounding body fluids upon fusion of multivesicular bodies and the plasma membrane. They were shown to carry cell-specific cargos of proteins, lipids, and genetic materials, and can be selectively taken up by neighboring or distant cells far from their release, reprogramming the recipient cells upon their bioactive compounds. Therefore, the regulated formation of exosomes, specific makeup of their cargo, cell-targeting specificity are of immense biological interest considering extremely high potential of exosomes as non-invasive diagnostic biomarkers, as well as therapeutic nanocarriers.

Induced pluripotent stem cells (iPSCs) are pluripotent stem cells generated from adult cells by reprogramming. iPSCs have the same properties as embryonic stem cells, and therefore self-renew and can differentiate into all cell types of the body except for cells in extra-embryonic tissues such as the placenta. iPSC-derived exosomes contain TGF- β、 BDNF etc., which can inhibit cell apoptosis, inhibit inflammatory response, promote angiogenesis, inhibit fibrosis, and enhance tissue repair potential, with a wide range of potential applications. iPSC-derived exosomes have emerged as an important paracrine factor for iPSCs to repair injured cells through the delivery of bioactive components.

The purpose of this trial is to evaluate the safety, tolerability, and preliminary efficacy of iPSC-derived exosomes in the treatment of atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years, body mass index (BMI) between 18 and 35 kg/m2 (including boundary values);
* Overall good health except AD;
* Participants diagnosed with atopic dermatitis (AD) as defined by the Hanifin and Rajka criteria;
* Investigator overall assessment (IGA) score of 2 to 3;
* Participants with a history of subacute or chronic AD symptoms for at least 6 months;
* Participants with body surface area (BSA) of AD involvement of ≤5% at screening and baseline;
* Participants and their partners agreed to use effective contraception throughout the study period (from screening to 3 months after completion of treatment);
* Participants understood and voluntarily signed the informed consent form.

Exclusion Criteria:

* There are obvious active systemic or local infections, including but not limited to the infection of AD secondary infection, local bacterial infection in target lesion, local viral infection in target lesion, and local fungal infection in target lesion. Note: After the infection resolves, the patients can be re-screened;
* Presence of any of the following conditions: HB surface antigen (HBsAg) positive and / or HB e antigen (HBeAg) positive, HB e antibody (HBeAb) and / or hepatitis B core antibody (HBcAb) positive and hepatitis B virus deoxyribonucleic acid (HBV-DNA) copy number> 2000 IU / mL; limited hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive; positive human immunodeficiency virus (HIV) antibody; positive for syphilis (TPA) test;
* Inoculate live or attenuated vaccine within 4 weeks before screening or during the study period;
* Received allergen specific immunotherapy within 6 months before screening;
* Use of topical drugs known or may affect AD within 2 weeks before screening (including but not limited to topical glucocorticoids; calcineurin inhibitors: such as tacrolimus, pirolimus, etc.);
* Use of immunosuppressants and Janus kinase inhibitors within 4 weeks before screening;
* Use of any biological agent (such as IL-4 receptor inhibitors, IL-13 inhibitors) for 12 weeks before screening or 5 half-lives (whichever is longer);
* Received systemic or local Chinese medicine treatment (including Chinese medicine immersion treatment) within 2 weeks before screening;
* Treated with UV and photochemistry within 4 weeks prior to screening;
* Required systemic treatment of antiviral, antiparasitic, antigenic, or antifungals within 4 weeks prior to screening;
* With significant abnormal findings or laboratory values and clinical significance, such as white blood cell count <3.0e9 / L; neutrophils <1 LLN; hemoglobin <90g / L; platelet <100e9 / L; serum creatinine> 1.5 ULN, ALT or AST 2 ULN; QTcF> 450 msec (male) or QTcF> 470 msec (female);
* Other combined (or co-occurrence) skin diseases that may affect the study evaluation, such as acne, psoriasis, lupus erythematosus, etc.; or large tattoos, birthmarks, skin scars, skin ulcers and other conditions that may affect the judgment of the investigator;
* Except for AD, any history of clinical major disease or clinically significant circulatory system abnormality, endocrine system abnormality, neurological or hematological disorders, immune system disease, psychiatric illness and metabolic instability; clinical significance is defined as the risk of the safety of the subject or aggravating the disease / disease during the study;
* Patients with a history of severe skin allergy and / or allergy to any ingredients of the product;
* History of cancer in the past 5 years (except for surgically removed squamous cell carcinoma, basal cell carcinoma, or skin carcinoma in situ);
* Any major surgery within 8 weeks before screening; or subjects expected to undergo surgery during the trial or within 4 weeks after the end of the trial; or 400 mL nonphysiological blood loss (including trauma, blood collection, blood donation within 12 weeks before screening);
* Pregnant women, lactating women, or women who plan to become pregnant during the study (fertile women must have a urine pregnancy test with negative results);
* Subjects who are currently participating in other clinical trials or who have participated in other clinical trials within 90 days;
* The investigator judged any other condition not suitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
adverse events as assessed by CTCAE | 42 days from post-administration
  all potentially treated subjects to assess the safety

SECONDARY OUTCOMES:
The proportion of subjects whose IGA score improved by 2 points or more compared with the baseline score. | Screening, after the first administration 8 day, 15 days, 21 days, 42 days
The proportion of subjects with an IGA score of 0-1 and an improvement of 2 or more over the baseline score | Screening, after the first administration 8 day, 15 days, 21 days, 42 days
The proportion of subjects whose EASI score improved by more than 50% compared with the baseline period | Screening, after the first administration 8 day, 15 days, 21 days, 42 days
The proportion of subjects whose EASI score improved by more than 75% compared with the baseline period | Screening, after the first administration 8 day, 15 days, 21 days, 42 days
The proportion of subjects whose EASI score improved by more than 90% compared with the baseline period | Screening, after the first administration 8 day, 15 days, 21 days, 42 days
Change in the score of the NRS | Screening, after the first administration 8 day, 15 days, 21 days, 42 days
Change in the score of the DLQI | Screening, after the first administration 8 day, 15 days, 21 days, 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhong Jin, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Science & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China